CLINICAL TRIAL: NCT02644590
Title: The Effect of Melatonin on Early Signs of Hypertension in Teenagers With Diabetes Mellitus Type 1
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Yonatan Yeshayahu, Dr, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 311080
Record Dates: First submitted 2015-12-28; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Type 1; Hypertension
Keywords: Melatonin; Nocturnal Hypertension; Type 1 Diabetes Melitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypertension | interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Melatonin treatment (Experimental): Adolescents with Type 1 Diabetes will undergo baseline 24 hour ambulatory blood pressure monitoring, followed by treatment with Melatonin for 3 weeks, using a single tablet at bed time, and repeat of the 24-hour blood pressure test following treatment period.
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — Detailed in arm description
  Other Names: Circadin

SUMMARY:
Nocturnal hypertension is recognized via ambulatory blood pressure monitoring in adolescents with type 1 diabetes mellitus.

Melatonin, (as previously seen in earlier studies in adults), may alter these changes, which may be a benefit especially for patients with diabetes mellitus who are at risk for cardiovascular changes.

The purpose of this study is to estimate the use of melatonin as treatment for nocturnal hypertension in young adults with type 1 diabetes melitus.

DETAILED DESCRIPTION:
Premature and extensive atherosclerosis and the increased risk for cardio-vascular disease (CVD) are the major causes of morbidity and mortality in patients with type 1 diabetes (T1DM), with an up to 20 fold increase in mortality from CVD . Most subjects with diabetes will develop hypertension which is a major determinant of both microvascular and cardiovascular complications.

The pediatric population is much less studied but nevertheless sufficient data suggest that the risk for CVD emerges during childhood. Up to 16% of adolescents with T1DM have hypertension, and studies using 24 hour ambulatory blood pressure monitoring (ABPM) in normotensive adolescents with T1DM have identified loss of diurnal systolic rhythm and nocturnal hypertension . Moreover, many normotensive patients, may have a loss of the physiologic drop in BP during the night ("non-dippers") and this too correlates with early vascular changes. This early change frequently leads to frank hypertension later on. The prevalence of CVD in this population points to the importance of early identification of known CVD risk factors and early intervention. Data from the Pathological Determinant in Youth (PDAY) study have shown that early changes leading to atherosclerosis exist in adolescence . These data stress the importance of identifying asymptomatic patients at the early stages of vascular changes.

Sleep and Hypertension:

During adolescence, total sleep duration changes and sleep/wake times shift such that teenagers go to bed late and wake up even later. The circadian timing system responsible for this phase delay in sleep is influenced by hormonal changes during puberty, specifically a delay in melatonin secretion . Only 20% of adolescents meet recommendations for hours of sleep during the week (9-9.25 h) , and adolescents frequently overcompensate on weekends with delayed awakening times . There is only limited data describing sleep patterns in type T1DM patients. Altered sleep may be of greater relevance in adolescents with T1DM, because disrupted sleep architecture occurs in children with diabetes, and sleep depravation does impair insulin sensitivity in diabetic subjects . We previously published a study comparing sleeping habits in diabetic and non-diabetic adolescents, showing that despite the intensive treatment they require which involves eating and injecting insulin at certain times, including in early morning, the diabetic adolescents did not make adjustments to their sleeping habits compared to healthy adolescents10. It has previously been reported that in certain situations where disrupted sleep occurs, including night shift workers, there is a loss of the "nocturnal dip" in blood pressure.11 In a preliminary observational study we performed in the diabetes clinic at Safra children's hospital we were able to identify more than 50% of adolescents with T1DM as "non-dippers" when measuring continuous BP using ABPM. More than 20% of diabetic adolescents had frank hypertension above the 95th %ile for age and height compared to 0% in the control group, and despite being normotensive during clinic visits12. In addition, a significant increase in hypertension load was seen in the diabetics compared to health controls only during sleep, and not wake hours.

All the information described above, points towards the hypothesis that adolescents with T1DM are at risk for developing nocturnal hypertension while still remaining normotensive when assessed during clinic visits.

Studies carried out by Grossman et al. at Sheba medical center showed impaired nocturnal melatonin secretion in non-dipper hypertensive patients, and improvement of nocturnal BP using controlled release (CR) melatonin. 13-14 Melatonin is a circulating neurohormone secreted predominantly at night. It is important in conveying the daily cycle of light and darkness to the body, thus regulating circadian rhythms. In addition to its' regulatory role, melatonin has antioxidative capacity, immunomodulatory potency, and anabolic properties that may be diminished by treatment with insulin. It has been shown that adolescents with T1DM secrete reduced levels of melatonin compared to healthy controls.15 Melatonin has been used for many years in the pediatric population for various sleep disorders and in studies assessing its other properties, including nocturnal BP control, and it has a good safety profile.16-17.

Study Aim:

To assess the effect of treatment with melatonin on nocturnal hypertension in adolescents and young adults with T1DM.

PROTOCOL DESCRIPTION

The suggested study will take place in the pediatric diabetes clinic at Sheba medical center. We aim to recruit 30 adolescents ages 12-21years T1DM. Recruitment phase is planned to last for a year.

Inclusion criteria: T1DM of at least 2 years. Exclusion criteria: 1. Known hypertension. 2. Use of BP lowering medication. 3. Abnormal kidney function or liver function. 4. Lactose intolerance.

Study design:

Cross sectional analysis: Each subject will have an overnight ABPM done. The purpose of this phase is to identify the subgroup of "non-dippers". The group of "non-dippers" will be recruited to the interventional phase.

Interventional phase: 15-20 subjects with an abnormal ABPM study will be treated with Melatonin-CR 2mg (Circadin®) for a total of 4 weeks and have a repeat of ABPM done. Comparison of ABPM results between the first test and the second test which is following 1 month of melatonin treatment will be done.

Methods:

Eligible patients will be approached and recruited during routine clinic visits. After consenting, the subjects will be provided with an ABMP device, either during clinic visits or delivered to their home by one of the investigators or research assistant. The patient will be instructed how to position the BP cuff on the arm and start the recording of BP. Blood pressure monitoring will be done using an ABPM device (SpaceLabs) which is commonly used for clinical purposes. During the following day after the test, the ABPM device will be collected from the family by the investigators.

Melatonin tablets will be provided to the subjects, and will be taken within 1 hour before they go to sleep at night. Subjects will be contacted following the first night of the study to monitor for adverse events, and the subjects will be provided with contact information of the researchers to report any adverse reactions that mey occur during the month of the study.

Safety:

Apart for the extensive use of melatonin in children, and an excellent safety profile, the specific brand used in this study - Circadin®, which is a controlled release formulation, has been used in multiple studies, including in children and has a good safety profile18-21.

Indications to termination of study participation of a participant:

1. Development of adverse effects to melatonin.
2. Intercurrent medical condition requiring hospitalization or treatment with BP lowering medication.
3. Participant or parents wish to stop the study for any reason.

Clinical surveillance during the study:

Participants will be contacted following the first night they receive melatonin and then weekly until completion of the study, to screen for adverse events. Participants will receive the direct phone number of a physician in the study group whom they can contact at any time with questions relating to the drug or adverse events during the study. Any adverse event will be documented and if severe, consideration will be give regarding stopping the study altogether with report to Helsinki committee and ministry of health.

Statistical analysis:

Rates of abnormal nocturnal BP will be compared between the pretreatment group and post treatment group using a x2 analysis. Continuous variables as systolic and diastolic BP will be compared using t-test, pre and post treatment.

Pearson's correlation coefficient will be used for correlation analysis between BP and clinical data as diabetes duration, metabolic control (HbA1c). Multivariate analysis will be used to assess clinical demographics which are strong predictors of nocturnal HTN.

Clinical importance:

Nocturnal hypertension as identified using ABPM is the earliest sign of hypertension in adolescents with T1DM. We have previously shown that it is present in a significant number of diabetic adolescents. Melatonin, as previously shown in adults, may modify these changes which would be a desirable effect in these patients at risk of cardiovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Teenagers and young adults with type 1 diabetes mellitus for at least two years

Exclusion Criteria:

* Previously known cardiovascular or renal disease
* Any previously use of antihypertensive drugs

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-09 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
blood pressure monitoring , pre and post treatment with melatonin | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yonatan Yeshayahu, MD, MHA, Principal Investigator — Sheba Medical Center